CLINICAL TRIAL: NCT00500279
Title: Effects of Celecoxib On Restenosis After Coronary Intervention and Evolution of Atherosclerosis Trial
Acronym: mini-COREA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-0611-011-188
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Last update posted 2007-07-12 (Estimated); Status verified 2007-07

CONDITIONS: Angioplasty, Transluminal, Percutaneous Coronary; Coronary Restenosis
Keywords: Drug-eluting stent; Restenosis; Celecoxib
MeSH Terms: conditions — Coronary Restenosis | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Celecoxib

SUMMARY:
To evaluate the effect of celecoxib use for 3 month after drug-eluting stent implantation

* on restenosis
* on clinical outcome such as target lesion revascularization, thrombotic event, myocardial infarction, death
* on inflammatory biomarkers

DETAILED DESCRIPTION:
Restenosis is the major adverse effect of coronary stent implantation. Drug-eluting stent has markedly reduced restenosis as compared with bare-metal stent, but restenosis is still the main cause of repeat coronary intervention after drug-eluting stent implantation. After coronary stent implantation, inflammatory reaction occurs in vessel wall and vascular smooth muscle cells proliferate. Celecoxib is well known to have anti-proliferative effect as well as anti-inflammatory effect, and safety of this drug is well-established. Celecoxib use for 6 month after paclitaxel-eluting stent implantation significantly reduced neointimal growth and repeat intervention without increase in adverse effect. Because inflammatory reaction seems to occur in very early period after vessel injury, reduced use of celecoxib may also be effective.

ELIGIBILITY:
Inclusion Criteria:

* angina pectoris or a positive stress test with native coronary artery lesions feasible for drug-eluting stent implantation

Exclusion Criteria:

* acute or recent ST segment elevation myocardial infarction (within four weeks)
* left main coronary artery disease
* hepatic dysfunction (AST or ALT > 120 IU/L )
* renal dysfunction (serum creatinine > 2.0 mg/dl)
* severe congestive heart failure (NYHA class > 2)
* left ventricular ejection fraction < 30%
* hemodynamically unstable condition
* definite intracoronary thrombus
* contraindication or history of allergy to aspirin, clopidogrel, or celecoxib
* warfarin use
* expected survival less than two years due to other medical conditions
* patients already taking any COX-3 inhibitor or NASIDS

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2006-11; Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
late luminal loss on quantitative coronary angiography | six month

SECONDARY OUTCOMES:
target lesion revascularization, myocardial infarction, death, thrombotic events | six and eighteen month

CONTACTS AND LOCATIONS:
Overall Officials: Hyosoo Kim, MD, PhD, Principal Investigator — Seoul National University Hospital; Bonkwon Koo, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam
  - Seuoul National University Hospital, Seoul

REFERENCES:
- [Background] Yang HM, Kim HS, Park KW, You HJ, Jeon SI, Youn SW, Kim SH, Oh BH, Lee MM, Park YB, Walsh K. Celecoxib, a cyclooxygenase-2 inhibitor, reduces neointimal hyperplasia through inhibition of Akt signaling. Circulation. 2004 Jul 20;110(3):301-8. doi: 10.1161/01.CIR.0000135467.43430.16. Epub 2004 Jul 6. PMID 15238462
- [Background] Wang K, Tarakji K, Zhou Z, Zhang M, Forudi F, Zhou X, Koki AT, Smith ME, Keller BT, Topol EJ, Lincoff AM, Penn MS. Celecoxib, a selective cyclooxygenase-2 inhibitor, decreases monocyte chemoattractant protein-1 expression and neointimal hyperplasia in the rabbit atherosclerotic balloon injury model. J Cardiovasc Pharmacol. 2005 Jan;45(1):61-7. doi: 10.1097/00005344-200501000-00011. PMID 15613981